CLINICAL TRIAL: NCT05844787
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study Including a Food Interaction Study, Followed by a Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability and Pharmacokinetics Profile of MT101-5 in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics Profile of MT101-5 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mthera Pharma Co., Ltd. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MT101-PD-001
Record Dates: First submitted 2023-03-07; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose (SAD) Study Including a Food Interaction Study, Followed by a Multiple Ascending Dose (MAD) Study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAD Phase (Experimental): SAD Phase: including Food Interaction - Blinding and Randomization: This is a randomized, double-blind, placebo-controlled, sentinel design, dose-escalating study with 40 healthy volunteers. Subjects will be assigned to 1 of up to 5 cohorts and will be randomized within each cohort to MT101-5 or placebo, as follows:
  * cohort 1: 100 mg (8 subjects total; 6 receiving MT101-5, 2 receiving placebo)
  * cohort 2: 150 mg (8 subjects total; 6 receiving MT101-5, 2 receiving placebo)
  * cohort 3: 300 mg (8 subjects total; 6 receiving MT101-5, 2 receiving placebo)
  * cohort 4: 450 mg (8 subjects total; 6 receiving MT101-5, 2 receiving placebo)
  * cohort 5: 600 mg (8 subjects total; 6 receiving MT101-5, 2 receiving placebo)
  Interventions: Drug: MT101-5
- Food Interaction Phase (Experimental): Food Interaction Phase: Following the completion of the SAD phase, if study stopping criteria (SSC) is not met, then subjects in cohort 5 will cross-over to the fed part of the study following a 7 day washout period. If SSC is achieved in the SAD phase, then the previous dose will be in the Food Interaction phase.
  Interventions: Drug: MT101-5
- MAD Phase (Experimental): MAD Phase; Blinding and Randomization: This is a randomized, double-blind, placebo-controlled study in approximately 8 elderly healthy volunteers. If study stopping criteria (SSC) is not met in the SAD phase, then subjects will be assigned to the cohort 5 dose. If SSC is achieved in the SAD phase, then the previous dose will be used as the cohort in the MAD phase
  Interventions: Drug: MT101-5

INTERVENTIONS:
Drug: MT101-5 — Tablet

SUMMARY:
The primary study objective is to establish the safety and tolerability of MT101-5 after a single and multiple dose administrations in healthy volunteers. The safety and overall tolerability of MT101-5 will be evaluated based on:

* Incidence of Dose Limiting Toxicities (DLTs)
* Incidence of Treatment-Emergent Adverse Events (TEAEs).
* Incidence of withdrawals due to Adverse Events (AEs).
* Change/shifts in laboratory values. Change in vital signs.
* Change in Electrocardiogram (ECG) parameters.
* Changes in physical examination findings

DETAILED DESCRIPTION:
SAD Phase including Food Interaction:

Subjects will be assigned to one of up to five MT101-5 treatment cohorts and will be randomly assigned 6:2 within their cohort to receive MT101-5 or placebo. On Day 1, following an overnight fast of at least 10 hours, the randomly assigned dose of MT101-5 or placebo will be administered as oral tablet in a fasting state with 240 mL (i.e., 8 fluid ounces) of water. Additional water is permitted ad lib except for the period 1 hour before to 1 hour after administration of the drug product. No food is allowed for at least 4 hours after the dose. Subjects should receive standardized meals scheduled at the same time throughout the study.

For the Food Interaction phase, on Day 1 following an overnight fast of at least 10 hours, the study subjects should start their standardized high-fat breakfast meal 30 minutes before administration of the drug product. Trial subjects should eat this meal in 30 minutes or less. Subjects will be administered MT101-5 or placebo as an oral tablet 30 minutes after start of intake of a standardized high-fat breakfast with 240 mL (8 fluid ounces) of water. Additional water is allowed ad lib except for 1 hour before and 1 hour after drug administration. No food is allowed for at least 4 hours after the dose.

MAD Phase:

Subjects will be randomly assigned 6:2 to receive MT101-5 or placebo once daily for 7 days. On Day 1, following an overnight fast of at least 10 hours, the randomly assigned dose of MT101-5 or placebo will be administered as oral tablet in a fasting state with 240 mL (i.e., 8 fluid ounces) of water. Additional water is permitted ad lib except for the period 1 hour before to 1 hour after administration of the drug product. No food is allowed for at least 4 hours after the dose. Subjects should receive standardized meals scheduled at the same time throughout the study. The same will be followed for days 2-7.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL of the following criteria:

1. Age:

   * SAD & Food Interaction: Healthy male and female subjects, 18 to 45 years of age, inclusive.
   * MAD: Elderly healthy male and female subjects ≥ 65 years of age
2. BMI:

   * SAD & Food Interaction: The subject has a body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, and weighs at least 50 kg.
   * MAD: The subject has a body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and weighs at least 50 kg.
3. The subject is in good health and has no medical condition of clinical significance or that may impact the outcome of the study, as determined by the investigator (as determined by medical history, physical examination, 12-lead electrocardiogram [ECG], vital signs, and clinical laboratory results at screening).
4. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
5. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
6. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided and has had the opportunity to discuss the study with the investigator or designee.
7. Negative pregnancy test for female subjects of childbearing potential. Women of childbearing potential (WOCBP) and Women of non-childbearing potential are eligible to participate. Both women of childbearing potential and women of non-childbearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 90 days after taking the last dose of MT101-5).

Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (e.g., diaphragm, cervical cap, male condom, and female condom and spermicidal foam, sponges, and film) (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile at least three months before screening (confirmed by study doctor) or 2 years post-menopausal (patient reported) confirmed with FSH/estradiol levels at screening. All male subjects/partners must agree to consistently and correctly use a condom for the duration of the study and for 90 days after taking the study drug. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.

Exclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet NONE of the following criteria:

1. The subject has a history of severe allergic or anaphylactic reactions.
2. The subject has a known allergy or hypersensitivity to any component of the formulation.
3. The subject has a medical history or current evidence of any clinically significant (as determined by the investigator) cardiac, endocrine (including diabetes), hematologic, hepatobiliary (abnormal alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transpeptidase [GGT], or total bilirubin), immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal condition, or other major disease.
4. The subject has a history of any malignant disease.
5. The subject has a history of more than one herpes zoster episode or multimetameric herpes zoster.
6. The subject has a history of an opportunistic infection (e.g. cytomegalovirus, pneumocystis carinii, aspergillosis, clostridium difficile).
7. The subject has a history of or ongoing chronic or recurrent infectious disease (e.g. infected indwelling prosthesis, osteomyelitis, chronic sinusitis).
8. The subject has had major trauma or surgery in the 2 months before screening or at any time between screening and check-in.
9. The subject has had an acute infection within 2 weeks before screening or at any time between screening and check-in including, but not limited to, history, signs, or symptoms of a common cold (e.g., mild rhinorrhea), untreated oral/dental abnormalities (e.g. untreated dental caries as determined by examination of the mouth), or untreated disruption of the skin.
10. The subject has clinically significant abnormal ECG findings at screening, check-in visits, or predose, as determined by the Investigator.
11. The subject has a supine blood pressure measurement outside the ranges of the below at screening, check-in, or predose. Note: If either value is out of the range, blood pressure measurements may be repeated in the supine position at intervals of 5 to 10 minutes up to 3 times. If the mean systolic or diastolic measurement continues to exceed the stated limits, the subject will be excluded.

    1. SAD: Ranges 90 to 140 mm Hg systolic or 45 to 90 mm Hg diastolic (measured after a rest of at least 5 minutes)
    2. MAD: Ranges 90 to 150 mm Hg systolic or 45 to 95 mm Hg diastolic (measured after a rest of at least 5 minutes)
12. The subject has a pulse of fewer than 45 beats per minute (bpm) or greater than 100 bpm (measured after a rest of at least 5 minutes) at screening, check-in, or predose.
13. The subject tests positive for tuberculosis (TB) at screening by the QuantiFERON-TB Gold Test, or has a history of latent, inadequately treated, or active TB.
14. The subject has a known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) types 1 or 2 at screening.
15. The subject has used prescription or over-the-counter (OTC) medication (other than ≤2 g/day paracetamol [acetaminophen] or ≤800 mg/day ibuprofen), vitamins, or herbal remedies, within 2 weeks or 5 half-lives before study drug administration, whichever is longer.
16. The subject has participated in another clinical study of a new investigational drug or has received an investigational drug within the 3 months or 5 half-lives (if available) before study drug administration, whichever is longer.
17. The subject has had a loss of more than 400 mL of blood (e.g. a blood donation) within 2 months before study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before check-in, or plans to donate blood during the study or within 3 months after the study.
18. The subject has a history of alcohol abuse (defined as an alcohol intake more than 21 units per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 240 mL of beer, 120 mL of wine, or 1 single shot of spirits. The subject will be required to abstain from alcohol consumption 48 hours prior to screening or check-in.
19. Current smokers and those who have smoked within the last 2 years. This includes the use of cigarettes, e-cigarettes, and nicotine replacement products.
20. The subject has a positive test for alcohol or drugs of abuse (barbiturates, methamphetamine, benzodiazepines, morphine/opiates, phencyclidine (PCP), amphetamines, tetrahydrocannabinol (THC), methylenedioxymethamphetamine (MDMA), cocaine, methadone, and cotinine) at screening or check-in.
21. The subject is unable to participate in, or successfully complete, the study, in the opinion of their general practitioner or the investigator, because the subject is any of the following:

    1. mentally or legally incapacitated, or unable to give consent for any reason
    2. in custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitarium or social institution
    3. unable to be contacted in case of emergency
    4. unlikely to cooperate or comply with the clinical study protocol or is unsuitable for any other reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Day 1 through 7 days after the last study drug administration
  Any clinically significant adverse event (AE)/serious adverse event (SAE) or clinically significant laboratory abnormality which is classified as > Grade 2 (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] version 5.0), where applicable, deemed by the investigator as at least "possibly, probably or definitely related" to the drug but unrelated to concurrent illness, or concomitant medications.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Day 1 through 7 days after the last study drug administration
  An adverse event (AE) is defined as any unfavorable or unintended sign, symptom, or disease that occurs or is reported by the patient to have occurred, or a worsening of a pre-existing condition. An adverse event may or may not be related to the study treatment.
Incidence of withdrawals due to Adverse Events (AEs) | Day 1 through 7 days after the last study drug administration
  Incidence of withdrawals due to Adverse Events (AEs) defined above
Change in complete blood count test | Change from baseline to day 7 after the first study drug administration
Change in comprehensive metabolic panel test | Change from baseline to day 7 after the first study drug administration
Change in urinalysis test | Change from baseline to day 7 after the first study drug administration
Change in pregnancy test | Change from baseline to day 7 after the first study drug administration
Change of blood pressure (both systolic and diastolic blood pressures) | Change from pre-dose to 96 hours after last study drug administration
Change of blood pressure (both systolic and diastolic blood pressures) | Change from pre-dose to day 7 after the last study drug administration
Change of pulse | Change from pre-dose to 96 hours after last study drug administration
Change of pulse | Change from pre-dose to day 7 after the last study drug administration
Change of temperature | Change from pre-dose to 96 hours after last study drug administration
Change of temperature | Change from pre-dose to day 7 after the last study drug administration
Change of respiratory rate | Change from pre-dose to 96 hours after last study drug administration
Change of respiratory rate | Change from pre-dose to day 7 after the last study drug administration
ECG ventricular rate (beats per minute) | At pre-dose
ECG ventricular rate (beats per minute) | 96 hours after study drug administration
ECG ventricular rate (beats per minute) | On day 7 after the last study drug administration
PR interval (msec) | At pre-dose
PR interval (msec) | 96 hours after study drug administration
PR interval (msec) | On day 7 after the last study drug administration
QRS interval (msec) | At pre-dose
QRS interval (msec) | 96 hours after study drug administration
QRS interval (msec) | On day 7 after the last study drug administration
QT interval (msec) | At pre-dose
QT interval (msec) | 96 hours after study drug administration
QT interval (msec) | On day 7 after the last study drug administration
QTc interval (msec) | At pre-dose
QTc interval (msec) | 96 hours after study drug administration
QTc interval (msec) | On day 7 after the last study drug administration
Maximum observed plasma drug concentration (Cmax) | 0-96 hours
Apparent terminal elimination half-life (t1/2) | 0-96 hours
Time to maximum observed plasma drug concentration (Tmax) | 0-96 hours
Area under the plasma drug concentration-time curve (AUC) | 0-96 hours
Percentage of AUC0-∞ extrapolated from Tlast to infinity (AUCext) | 0-96 hours
Apparent plasma clearance (CL/F) | 0-96 hours
Apparent Volume of distribution (Vz/F) | 0-96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services, 1nc., Secaucus, New Jersey, United States